CLINICAL TRIAL: NCT04178525
Title: A Randomized, Parallel, Double Blind, Placebo Controlled, Multicentre, Two Arms Clinical Trial Evaluating the Safety and Efficacy of the Use of Chitosan Gel in Patients With Chronic Wounds
Brief Title: Clinical Trial Evaluating the Safety and Efficacy of the Use of Chitosan Gel in Patients With Chronic Wounds
Acronym: CHITOWOUND
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 restrictions
Sponsor: Primex ehf (Industry)
Collaborators: Vizera d.o.o. (Industry); University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHITO-01
Record Dates: First submitted 2019-11-13; First posted 2019-11-26 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Diabetic Foot Ulcer
Keywords: Chronic wounds; Diabetic foot ulcer; Chitosan gel
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Randomization will be applied at a 1:1 ratio on study level, and at each individual site. Sixty (60) patients will be included in the study, 30 in each arm.
Who Masked: Participant, Investigator
Masking Description: The patients, investigators and other personnel involved in the study will be blinded with respect to the study treatment of the patient, until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental group (Experimental): ChitoCare gel administered topically 2-3 times a week or more (accordingly with the frequency of dressing change)
  Interventions: Device: ChitoCare gel
- Arm B (Control group) (Placebo Comparator): Placebo gel administered topically 2-3 times a week or more (accordingly with the frequency of dressing change)
  Interventions: Device: Placebo gel

INTERVENTIONS:
Device: ChitoCare gel — ChitoCare gel is based on chitosan and used as an addition to standard care, accordingly with dressing change for 10 weeks.
  Arms: Arm A (Experimental group
Device: Placebo gel — Placebo gel is used as an addition to standard care, accordingly with dressing change for 10 weeks.
  Arms: Arm B (Control group)

SUMMARY:
Type 1 and Type 2 diabetic patients with diabetic foot ulcer will be recruited and screened for participation in the study. Eligible patients will be randomized 1:1 to either experimental or control group and undergo 10-weeks of treatment (as an addition to standard care) and 4 weeks of follow-up to evaluate the effect of chitosan gel on chronic wound (diabetic foot ulcer) healing.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be given
* Patient ≥ 18 years old
* Diagnosed with type I or type II diabetes mellitus
* Glycosylated haemoglobin, HbA1c, ≤ 12%
* Presence of diabetic foot ulcer or an amputation wound that meets following criteria:

  1. Size of the wound 0,5 - 12 cm^2
  2. Wagner grade I or II
  3. Wound is not infected
  4. Wound present for at least 4 weeks
* If multiple wounds are present, the biggest wound fitting the criteria is selected and the distance from other wounds must be at least 2 cm
* If there is an amputation wound present, it can be used for the purpose of this study if it fits the rest of the criteria
* Adequate perfusion (good, strong foot pulses). If foot pulses are weak, evaluation of perfusion pressures with Doppler ultrasound is performed.
* Able to understand and comply with the requirements of the trial

Exclusion Criteria:

* Known history of alcohol or drug abuse
* Use of any antibiotic medication within the last 7 days prior to the first application of study product
* Patients presenting with Wagner Grade III or higher ulcer
* Patients with serious concomitant disease (cancer, heart failure ( NYHA class IV), severe anemia (Hb<100 g/L), neoplasia)
* Any significant condition that may preclude the participant from the study (e.g. severe depression or psychiatric illness)
* Patients that will require surgical procedure to treat their ischemic condition on the limb where the wound is present as assessed by the doctor
* Excessive lymphedema that could interfere with wound healing (if there is mild edema treated with compression therapy the patient can be included)
* Patients diagnosed with autoimmune connective tissues diseases
* Previous treatment under this clinical protocol
* Participation in another clinical trial up to 30 days before the randomization visit.
* Receiving or scheduled to receive a medication or treatment which, in the opinion of the investigator, was known to interfere with, or affect the rate and quality of wound healing
* Medical condition likely to require systemic corticosteroids during the study period
* Allergic to shellfish, chitosan or one of ChitoCare product compounds
* Immobile patients
* Pregnant and lactating women
* Significant increase in wound healing during run-in period (reduction of wound size area ≥ 40%)
* BMI > 39 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Difference in proportions of ulcers completely healed for experimental group compared to control group. | 10 weeks
  Relative healing rate (ratio between the proportion of ulcers healed for experimental group to proportion of ulcers healed in control group (= healing rate)).

SECONDARY OUTCOMES:
Difference in proportion of ulcers completely healed for experimental group compared to the control group | 2, 4, 6 and 8 weeks
  Relative healing rate (ratio between the proportion of ulcers healed for experimental group to the proportion of ulcers healed in control group)
Difference in reduction of diabetic ulcer wound size for experimental group compared to control group. | 2, 4, 6, 8, 10 and 14 weeks
  Relative reduction of wound surface area.
Difference in time to complete healing for experimental group compared to control group. | Baseline to 14 weeks (whole study duration)
  Hazard ratio for time to complete healing (experimental group vs. control group)
Difference in improved quality of life for experimental group compared to control group. | 4 weeks and 10 weeks
  The relative improvement of quality of life from the baseline value using the 36-Item Short Form Survey (SF-36) questionnaire (RAND Corporation).
Difference in improved state of the wound for experimental group compared to control group using Bates-Jensen wound assessment tool (BWAT). | 2, 4, 6, 8, 10 and 14 weeks
  The relative improvement of the state of the wound using Bates-Jensen wound assessment tool (BWAT).
Difference in improved state of the wound for experimental group compared to control group according to Wagner Ulcer Classification. | 2, 4, 6, 8, 10 and 14 weeks
  The relative improvement of the state of the wound using Wagner Ulcer Classification.
Secondary infections that may occur during the study for experimental group compared to control group. | Baseline to 14 weeks (whole study duration)
  Occurrence of secondary infection.
Incidence of treatment related adverse events for experimental group compared to control group. | Baseline to 14 weeks (whole study duration)
  The incidence of treatment related adverse events.
To track diabetic ulcer recurrence for experimental group compared to control group in patients whose wound completely healed. | Baseline to 14 weeks (whole study duration)
  The incidence of diabetic ulcer recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Maja Navodnik Preložnik, MD, Principal Investigator — General Hospital Celje, Slovenia
Locations (5):
- University Clinic Vuk Vrhovac, Zagreb, Croatia
- Slovenia (4):
  - General Hospital Celje, Celje
  - Clinic Golnik - Diabetic Clinic Kranj, Kranj
  - University Hospital Center Ljubljana, Ljubljana
  - General Hospital Murska Sobota, Murska Sobota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Slivnik M, Navodnik Preloznik M, Fir M, Jazbar J, Cebron Lipovec N, Locatelli I, Liette Lauzon H, Urbancic Rovan V. A randomized, placebo-controlled study of chitosan gel for the treatment of chronic diabetic foot ulcers (the CHITOWOUND study). BMJ Open Diabetes Res Care. 2024 Jun 23;12(3):e004195. doi: 10.1136/bmjdrc-2024-004195. PMID 38909998